CLINICAL TRIAL: NCT00113997
Title: The Healthy Volunteer Evaluation of an Aptamer-RNA Target to Factor IXa
Brief Title: Safety and Dosing Evaluation of REG1 Anticoagulation System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050164; 05-H-0164
Record Dates: First submitted 2005-06-11; First posted 2005-06-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Healthy
Keywords: Anticoagulant; Antidote; Pharmacokinetics; Pharmacodynamics; Healthy Volunteer; HV

INTERVENTIONS:
Drug: REG1

SUMMARY:
This 1-week study will test the safety and dosing of an anticoagulation system called REG1 that is designed to improve control of "blood thinning." Patients with heart attack and other conditions require treatment with an anticoagulant (blood thinner) to prevent the formation of blood clots. However, anticoagulation therapy can increase the risk of bleeding. The REG1 system is designed to minimize this risk. One part of the system stops the activity of factor IX (a protein that helps blood clot) while the other part of the system (the antidote) inactivates the drug and stops the thinning process. This study will examine in normal healthy subjects how the REG1 system works in the body and how it leaves the body.

Healthy normal volunteers between 12 and 65 years of age who weigh 50-120 kilograms (110-264 pounds) and have no history of bleeding problems or significant bleeding may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood tests.

Participants must avoid foods that may alter the blood's clotting ability and must not take any medications the week of the study. They undergo the following tests and procedures:

Day 1

Subjects are admitted to the NIH Clinical Center for an overnight stay. Two catheters (plastic tubes) are placed in the subject's arm veins, one for drawing blood samples and the other for injecting one of the following: REG1 drug, REG1 antidote, REG1 drug and antidote, or placebo. Two injections of study medication are given, spaced 3 hours apart, each over a 1-minute period. After each injection, blood is collected at specific times to measure levels of the drug or antidote in the body and the blood's ability to clot. Subjects also provide a 24-hour urine collection and stool sample.

Day 2

A blood sample is drawn 24 hours after the drug or antidote injection from the previous day. If the blood test result is normal, subjects are discharged home with instructions to follow. They return to the Clinical Center at 36 hours and 48 hours for additional blood samples.

Days 3 and 7

A blood sample is collected at the end of day 3 and day 7. Urine and stool samples are also collected.

DETAILED DESCRIPTION:
Given the central role of thrombosis in the pathobiology of acute ischemic heart disease, injectable (intravenous or subcutaneous) anticoagulants have become the foundation of medical treatment for patients presenting with acute coronary syndromes (unstable angina and myocardial infarction; ACS) and for those undergoing coronary revascularization procedures, either percutaneously or surgically (Harrington et al., 2004; Popma et al., 2004). Currently available anticoagulants include unfractionated heparin (UFH), the low molecular weight heparins (LMWH), and the direct thrombin inhibitors (DTI) (e.g., recombinant hirudin, bivalirudin, and argatroban). The present paradigm both for anticoagulant use and for continued antithrombotic drug development is to establish a balance between efficacy (reducing the risk of ischemic events) and safety (minimizing the risk of bleeding) (Harrington et al., 2004). Each of the available agents carries an increased risk of bleeding relative to placebo.

The major adverse event associated with anticoagulant and antithrombotic drugs is bleeding, which can cause permanent disability and death (Ebbesen et al., 2001; Levine et al., 2004). Generally, cardiovascular clinicians have been willing to trade off an increased risk of bleeding when a drug can reduce the ischemic complications of either the acute coronary syndromes or of coronary revascularization procedures. However, recent data have suggested that bleeding events, particularly those that require blood transfusion, have a significant impact on the outcome and cost of treatment of patients with ACS. Transfusion rates in patients undergoing elective coronary artery bypass graft (CABG) surgery range from 30-60%, and transfusion in these patients is associated with increased short, medium and long-term mortality (Bracey et al., 1999; Engoren et al., 2002; Hebert et al., 1999). Bleeding is also the most frequent and costly complication associated with percutaneous coronary interventions (PCI), with transfusions being performed in 5-10% of patients at an incremental cost of $8000-$12,000 (Moscucci, 2002). In addition, the frequency of significant bleeding in patients undergoing treatment for ACS is high as well, ranging from 5% to 10% (excluding patients who undergo CABG), with bleeding and transfusion independently associated with a significant increase in short-term mortality (Moscucci et al., 2003; Rao et al., 2004). Therefore, despite the continued development of novel antithrombotics, a significant clinical need exists for safer anticoagulant agents.

For hospitalized patients with acute ischemic heart disease, the ideal anticoagulant would be deliverable by intravenous or subcutaneous injection, immediately effective, easily dosed so as not to require frequent monitoring and immediately and predictably reversible.

UFH is the only antidote-reversible anticoagulant currently approved for use. However, UFH has significant limitations. First, heparin has complex pharmacokinetics that make the predictability of its use challenging (Granger et al., 1996). Second, the dose predictability of its antidote, protamine, is challenging, and there are serious side effects associated with its use (Carr and Silverman, 1999; Welsby et al., 2005). Finally, heparin can induce thrombocytopenia (HIT) and thrombocytopenia with thrombosis (HITT) (Warkentin, 2005; Warkentin and Greinacher, 2004).

Despite these limitations, heparin remains the most commonly used anticoagulant for hospitalized patients primarily because it is "reversible." Newer-generation anticoagulants, such as the LMWHs have improved upon the predictability of UFH dosing and do not require lab-based monitoring as part of their routine use. HIT and HITT are observed less frequently with the LMWHs, relative to UFH, but they have not eliminated this risk. Two of the three commercially available DTIs, lepirudin and argatroban, are specifically approved for use in patients who have developed or have a history of HIT. Bivalirudin is approved for use as an anticoagulant during PCI and therefore provides an attractive alternative to UFH in patients who have HIT. However, there are no direct and clear antidotes to reverse the anticoagulant effects of the LMWHs, nor of the DTIs, which presents a particular risk to their use in patients undergoing surgical or percutaneous coronary revascularization procedures (Jones et al., 2002). Bleeding in patients treated with LMWH's or DTI's is managed by administering blood products (including clotting factor).

Rapid reversal of drug activity can be achieved by formulation of a drug as an infusible agent with a short half-life, or via administration of a second agent, an antidote, that can neutralize the activity of the drug. Short-acting direct thrombin inhibitors such as bivalirudin, which can be reversed simply by cessation of infusion, are being developed as infusible anticoagulants for use in CABG surgery (Merry et al., 2004). However, the co-morbidities such as renal dysfunction, present in a large percentage of patients undergoing CABG (or PCI) procedures (Al Suwaidi et al., 2002), may preclude rapid clearance of the drug and thus delay reversal of activity, and/or the relatively large quantity of drug required to sustain anticoagulation (i.e., necessary to achieve effective steady state levels of a short-half-life agent) may significantly interact with underlying renal impairment to compound the problem. Therefore, it remains to be seen if these drugs will indeed achieve rapid reversal of anticoagulation following stoppage of infusion in the target patient populations, and whether the clearance of the drug itself may exacerbate renal dysfunction.

An alternative approach to providing controlled anticoagulation embraced by Regado Biosciences is the utilization of an anticoagulating agent with medium-term duration of action (~12 hours) that can achieve clinically appropriate activity at relatively low doses, in combination with a second agent capable of specifically binding to and neutralizing the primary anticoagulant. Such a "drug-antidote" combination can ensure predictable and safe neutralization and reversal of the anticoagulant activity of the drug (Rusconi et al., 2004; Rusconi et al., 2002).

The cell-based model of coagulation (Hoffman et al., 1995; Kjalke et al., 1998; Monroe et al., 1996) (Figure 1) provides the clearest explanation to date of how physiologic coagulation occurs in vivo. The advance of this model over prior descriptions of the coagulation reaction is that it incorporates the cellular surfaces upon which the specific coagulation factors accumulate and react, and thereby more accurately explains the phenotypes observed in individuals lacking, or deficient in, the various coagulation factors and platelet receptors.

According to this model, the procoagulant reaction occurs in three distinct steps, initiation, amplification and propagation. Initiation of coagulation takes place on tissue factor-bearing cells (e.g., activated monocytes, macrophages, and endothelial cells). Coagulation factor VIIa, which forms a complex with tissue factor, catalyzes the activation of coagulation factors IX (FIX) and X (FX), which in turn generates a small amount of thrombin from prothrombin. In the amplification phase (also referred to as the priming phase), the small amount of thrombin generated in the initiation phase activates coagulation factors V, VIII, and XI and also activates platelets, which supplies a surface upon which further procoagulant reactions occur. In vivo, the small amounts of thrombin generated during the amplification phase are not sufficient to convert fibrinogen to fibrin, due to the presence of endogenous thrombin inhibitors termed serpins, such as anti-thrombin III, -2-macroglobulin and heparin cofactor II. The final phase of the procoagulant reaction, propagation, occurs exclusively on the surface of activated platelets. During propagation, significant amounts of FIXa are generated by the FXIa-catalyzed activation of FIX. FIXa forms a complex with its requisite cofactor FVIIIa, which activates FX. Subsequently, FXa forms a complex with its requisite cofactor FVa. The FXa-FVa complex activates prothrombin, which leads to a "burst" of thrombin generation and fibrin deposition. The end result is the formation of a stable clot.

Based upon this model, FIXa play two roles in coagulation. In the initiation phase, FIXa plays an important role in generating small amounts of thrombin via activation of FX to FXa and subsequent prothrombin activation. However, this role of FIXa is at least partially redundant with the tissue factor FVIIa-catalyzed conversion of FX to FXa. The more critical role of FIXa occurs in the propagation phase, in which the FVIIIa/FIXa enzyme complex serves as the sole catalyst of FXa generation on the activated platelet surface. Therefore, a reduction in FIXa activity, either due to genetic deficiency in FIX (i.e. hemophilia B) or pharmacologic inhibition of FIX/IXa, is expected to have several effects on coagulation. First, inhibition or loss of FIXa activity should partially dampen the initiation of coagulation. Second, inhibition or loss of FIXa activity should have a profound effect on the propagation phase of coagulation, resulting in a significant reduction or elimination of thrombin production. Finally, limitation of thrombin generation during the propagation phase will at least partially quell feedback amplification of coagulation by reducing activation of platelets and upstream coagulation factors such as factors V, VIII and XI.

Inhibitors of FIX activity, such as active site-inactivated factor IXa (FIXai) or monoclonal antibodies against FIX (e.g., the antibody BC2), have exhibited potent anticoagulant and antithrombotic activity in multiple animal models, including various animal models of arterial thrombosis and stroke (Benedict et al., 1991; Choudhri et al., 1999; Feuerstein et al., 1999; Spanier et al., 1998a; Spanier et al., 1997; Spanier et al., 1998b; Toomey et al., 2000). In general, these studies have shown that FIXa inhibitors have a higher ratio of antithrombotic activity to bleeding risk than unfractionated heparin in animals. However, in these studies, at doses marginally higher than the effective dose, animals treated with these agents have exhibited bleeding profiles no different than heparin. Such an experience in well-controlled animal studies suggests that, in the clinical setting, the ability to control the activity of a FIXa inhibitor would enhance its safety and facilitate its medical use. In addition, FIXai has been shown to be safe and effective as a heparin replacement in multiple animal surgical models requiring anticoagulant therapy, including rabbit models of synthetic patch vascular repair, as well as canine and non-human primate models of CABG with cardiopulmonary bypass (Spanier et al., 1998a; Spanier et al., 1997; Spanier et al., 1998b). FIXai has also been used successfully for several critically ill patients requiring cardiopulmonary bypass and in the setting of other extracorporeal circuits such as extracorporeal membrane oxygenation (Spanier et al., 1998a) by physicians at the Columbia College of Physicians and Surgeons, on a compassionate care basis. Thus, FIXa is a validated target for anticoagulant therapy in coronary revascularization procedures (both CABG and PCI), and for the treatment and prevention of thrombosis in patients suffering from acute coronary syndromes.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants are eligible if they meet the following criteria:
* Age is greater than or equal to 21 years to 65 years
* Ability to give written informed consent
* Weight between 50 Kg and 120 Kg

EXCLUSION CRITERIA:

* Participants are NOT eligible under the following conditions:
* Age is less than 21 years
* Subject weight is less than 50 Kg of greater than 120 Kg
* Females - Pregnant or lactating
* Females - active menstruation on day of injection (Females may be randomized if they are not actively menstruating on day of injection or they can be randomized as soon as menstruation ceases)
* Any medical condition (other than a self-limited illness) that requires ongoing and current medical attention
* Any prescription medication (including oral or patch or injectable contraceptives)
* Any use of NSAIDS or aspirin in the prior 7 days
* Any known individual or family history of a bleeding diathesis or coagulopathy
* Any history of thrombocytopenia, or baseline platelet count less than 150,000
* Any history of thrombocytosis or baseline platelet count greater than 600,000
* Endoscopic peptic ulcer disease in the past 3 years or GI bleeding in the past 3 months
* Genitourinary bleeding within the past 3 months
* Severe trauma, fracture, major surgery, or biopsy of a parenchymal organ within the past 3 months
* Any evidence or history of intracranial bleeding or aneurysm
* Any history of thrombotic or hemorrhagic stroke
* Severe persistent hypertension (systolic pressure greater than 180 mm Hg or diastolic greater than 110 mm Hg)
* Baseline Hgb less than 12.0 g/dL, PT greater than ULN, or APTT greater than ULN
* Baseline liver dysfunction (ALT, AST, bilirubin, or alkaline phosphatase greater than ULN)
* Baseline renal dysfunction (serum creatinine or BUN greater than ULN)
* Use of an investigational drug within the past 30 days
* Any factor that might influence ability to return for follow-up visits
* Illicit drug or alcohol abuse
* Inability to comply with the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106
Dates: Start 2005-06; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Al Suwaidi J, Reddan DN, Williams K, Pieper KS, Harrington RA, Califf RM, Granger CB, Ohman EM, Holmes DR Jr; GUSTO-IIb, GUSTO-III, PURSUIT. Global Use of Strategies to Open Occluded Coronary Arteries. Platelet Glycoprotein IIb/IIIa in Unstable Angina: Receptor Suppression Using Integrilin Therapy; PARAGON-A Investigators. Platelet IIb/IIIa Antagonism for the Reduction of Acute coronary syndrome events in a Global Organization Network. Prognostic implications of abnormalities in renal function in patients with acute coronary syndromes. Circulation. 2002 Aug 20;106(8):974-80. doi: 10.1161/01.cir.0000027560.41358.b3. PMID 12186803
- [Background] Benedict CR, Ryan J, Wolitzky B, Ramos R, Gerlach M, Tijburg P, Stern D. Active site-blocked factor IXa prevents intravascular thrombus formation in the coronary vasculature without inhibiting extravascular coagulation in a canine thrombosis model. J Clin Invest. 1991 Nov;88(5):1760-5. doi: 10.1172/JCI115495. PMID 1939660
- [Background] Bracey AW, Radovancevic R, Riggs SA, Houston S, Cozart H, Vaughn WK, Radovancevic B, McAllister HA Jr, Cooley DA. Lowering the hemoglobin threshold for transfusion in coronary artery bypass procedures: effect on patient outcome. Transfusion. 1999 Oct;39(10):1070-7. doi: 10.1046/j.1537-2995.1999.39101070.x. PMID 10532600